# **Allegro Evaluation Protocols**

Nova Biomedical | Medical & Scientific Affairs

Version 3: 18 July 2016

# **Preface**

Clinical laboratory based method evaluations are a set of studies aimed at characterizing the performance of an assay – a procedure for qualitatively assessing or quantitatively measuring the presence or amount of a target entity, i.e. analyte or measurand. These studies utilize controlled experimental technique to assess the various components of a measurement including the assessment of: method comparison, reproducibility, specificity, and accuracy. Highly accurate and precise measurements are central to the practice of laboratory medicine given that these measurements are used to manage the patient throughout the entire spectrum of care. It is therefore necessary that clinical laboratorians perform their due diligence in the careful selection and subsequent management of laboratory methods. In order to assist the investigator, a collection of evaluation protocols specifically designed to assess the performance of the Allegro has been provided. These protocols are based on the recommendations provided by the Clinical and Laboratory Standards Institute (CLSI), a recognized body that publishes consensus guidelines on the various practice aspects of laboratory medicine.

# Introduction

Allegro is a fast, simple, capillary whole blood analyser with a diabetes-focused menu.

The comprehensive test menu available on the Allegro is:

Glycemic Control Lipid Kidney Function

HbA1c Total Cholesterol Urine Creatinine

HDL Cholesterol Urine Albumin

Triglyceride

The Allegro can be used in conjunction with the companion tests below to further extend the diabetes management menu

# **Companion Tests**

Anemia – Hemoglobin and Hematocrit Glycemic control – Glucose and Ketone

**HbA1c, Lipid and Kidney Function tests** are provided in their own multi test cartridge so each cartridge measures all analytes within each profile

# Scope

The scope of this protocol is to evaluate and assess the analytical performance of the HbA1c, Lipid cartridge and the Kidney Function cartridge.

Analytical performance will be assessed on each profile e.g. Lipid, HbA1c, and Kidney Function, independently and will comprise of:

Within Day precision
Between Day precision
Method Correlation

## **Supplemental System Specifications:**

# **Operating Environment:**

Operating Location:

The analyzer is intended for indoor operation on a stationary, stable, bench.

Operating Temperature and Relative Humidity Range:

The Analyzer shall be able to operate under the following conditions

Operating Temperature Range: 15 to 32°C (59°F to 90°F)
 Relative Humidity Range: 20 – 85%, non-condensing

Altitude:

The Analyzer shall be able to operate at an altitude of up to 3,660 meters (12,000 feet)

# **Power Requirements:**

Operating Voltage: 90 to 264 VAC

Operating Frequency: 50/60Hz

# **Contents**

# 1. Kidney Function (Tests: Urine Creatinine and Albumin)

- I. Within Day Precision Study Protocol
- II. Between Day Precision Study Protocol
- III. Method Comparison Protocol
- IV. Summary Report Template

# 2. Glycemic Control (Tests: HbA1c)

- I. Within Day Precision Study Protocol
- II. Between Day Precision Study Protocol
- III. Method Comparison Study Protocol
- IV. Summary Report Template

# 3. Lipid (Tests: Total Cholesterol, Triglycerides, HDL Cholesterol

- I. Within Day Precision Study Protocol
- II. Between Day Precision Study Protocol
- III. Method Comparison Study Protocol
- IV. Summary Report Template

# 1. Urine Creatinine and Albumin

I. Within Day Precision Study Protocol

Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

# **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the within day precision of urine creatinine and urine Albumin measurements on the Allegro system.

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Kidney Function Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic tubes for decanting urine samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

# **Important Factors to Consider**

Tests: Urine Creatinine and Urine Albumin

Sample Type: Fresh random urine

**Sample Size:** 25μL **Time per UACR:** 7 mins

**Linear Range of Operation:** 15-500 mg/dL (13.0-44.2 mmol/L) **Linear Range of Operation for urine Albumin:** 5-300 mg/L

# **Expected Normal Values**

Urine Creatinine: For a random urine sample, >12 Years Male 20-370 mg/dL (1.8- 32.7 mmol/L), >12 Years

Female 20 – 320 mg/dL (1.8-28.3 mmol/L)

**Urine Albumin:** For a random urine sample, normal values are typically 0 to 30 mg/L

#### **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

**Urine Albumin and Creatinine:** 

Low Level Target: Urine Albumin ~50 mg/L Creatinine ~85 mg/dL (~8 mmol/L)

High Level Target: Urine Albumin ~180 mg/L Creatinine ~220 mg/dL (~20 mmol/L)

Please note that urine creatinine and Albumin are processed at the same time and can be run in both channels.

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. Select low, med and high levels of both urine creatinine and Albumin, ideally using discarded random urine collections or, if these are not available, then urine samples that have been spiked with appropriate concentrations of creatinine spiking solution and/or human Albumin (may need to be tested for homogeneity).
- 4. Suggested concentrations for low, medium and high samples: -

- 5. Ensure adequate mixing before analysis.
- 6. Cartridges are stored at 4° each cartridge requires 10-15 mins warm up time so consider this requirement when planning study needs.
- 7. Run each Level <u>10</u> times on Allegro, consider running only in one channel to reduce variability. Record results on Data Collection Sheet.
- 8. Total Analysis Time:  $7 \text{ mins } x \cdot 10 = 70 \text{ mins per level}$ . 210 mins for all levels. Approx. 3.5 hrs plus preparation time.

## **Data Analysis**

The within-run precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1].

#### **Data Review**

This data will be summarized in a final report which will also include an assessment of the accuracy. This report should be reviewed by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of Allegro performance prior to the conductance of clinical studies.

# References

| 1. | Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative |
|---|---|
| | Measurement Methods; Approved Guideline – Second Edition. EP5-A2. |

# Appendix 1

# Within-Day Precision Study Data Collection Sheet

| Hospital Name: | Date of Study: |
|------------------------------------|---------------------------|
| System Operator(s): | |
| Reference Analyzer | |
| Level 1 Urine Creatinine and Urine | <u>Albumin</u> |
| Reference Analyzer Result: Urine C | reatinine mg/dL or mmol/L |
| Reference Analyzer Result: Urine A | llbumin mg/L or g/L |

| | System Name | | |
|---|---|---|---|
| | System Serial # | | |
| | Cartridge Lot # | | |
| Low QC | Range: | | |
| High QC | Range: | | |
| | Replicate # | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Albumin<br>Result<br>mg/L or g/L |
| | 1 | | |
| | 2 | | |
| | 3 | | |
| | 4 | | |
| | 5 | | |
| | 6 | | |
| | 7 | | |
| | 8 | | |
| | 9 | | |
| | 10 | | |

# Level 2 Urine Creatinine and Urine Albumin

| Reference Analyzer Result: Urine Creatinine mg/dL or mmol/L |
|-------------------------------------------------------------|
| Reference Analyzer Result: Urine Albumin mg/L or g/L |

| | System Name | | | |
|---|---|---|---|---|
| | System Serial # | | | |
| | Cartridge Lot # | | | |
| Low QC | Range: | | | |
| High QC | Range: | | | |
| | Replicate # | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Albumin<br>Result<br>mg/L or g/L | |
| | 1 | | | |
| | 2 | | | |
| | 3 | | | |
| | 4 | | | |
| | 5 | | | |
| | 6 | | | |
| | 7 | | | |
| | 8 | | | |
| | 9 | | | |
| | 10 | | - | - |

# Level 3 Urine Creatinine and Urine Albumin

| Reference Analyzer Result: Urine Creatinine mg/dL or mmol/L |
|-------------------------------------------------------------|
| Reference Analyzer Result: Urine Albumin mg/L or g/L |

| | System Name | | |
|---|---|---|---|
| | System Serial # | | |
| | Cart Lot # | | |
| Low QC | Range: | | |
| High QC | Range: | | |
| | Replicate # | Urine Creat<br>Result mg/dL or<br>mmol/L | Urine Albumin<br>Result<br>mg/L or g/L |
| | 1 | | |
| | 2 | | |
| | 3 | | |
| | 4 | | |
| | 5 | | |
| | 6 | | |
| | 7 | | |
| | 8 | | |
| | 9 | | |
| | 10 | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |

| I. Urine Creatinine and Urine Albumin |
|------------------------------------------|
| II. Between-Day Precision Study Protocol |

Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). *Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition.* EP5-A2.

# **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the between-day precision of urine creatinine and urine Albumin measurements on the Allegro system.

### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Kidney Function Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic tubes for decanting urine samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

# **Important Factors to Consider**

Tests: Urine Creatinine and Urine Albumin

Sample Type: Fresh random urine

Sample Size: 25μL Time per UABCR: 7 mins

Linear Range of Operation for Urine Creatinine: 15-500 mg/dL (13.0-44.2 mmol/L)

Linear Range of Operation for Urine Albumin: 3-300 mg/L

#### **Expected Normal Values**

Urine Creatinine: For a random urine sample, >12 Years Male 20-370 mg/dL (1.8- 32.7 mmol/L), >12 Years

Female 20 – 320 mg/dL (1.8-28.3 mmol/L)

Urine Albumin: For a random urine sample, normal values are typically 0 to 30 mg/dL

# **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

**Urine Albumin and Creatinine:** 

Low Level Target: Urine Albumin ~50 mg/L Creatinine ~85 mg/L (~8 mmol/L)

High Level Target: Urine Albumin ~180 mg/L Creatinine ~220 mg/L (~20 mmol/L)

Please note that urine creatinine and urine Albumin are processed at the same time

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Analyse controls on Allegro every day that testing is carried out, 2 runs per day would be performed one in the morning and the other in the afternoon so QC would need to be performed prior to each run, make sure results are within specification before proceeding. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. Select low, med and high levels of both urine creatinine and Albumin. These can be obtained from one or more of the following: a) samples from random urine collections, b) samples spiked with stock concentrations of Albumin and/or creatinine, or c) samples used for the within day precision test. Forty aliquots must be prepared from each sample and frozen.
- 4. A freshly thawed aliquot will then be analysed every morning and afternoon in duplicate for 10 consecutive working days
- 5. Suggested concentrations for low, medium and high samples: -

| | Urine Creatinine | Urine Albumin |
|---------------|-------------------------------|-------------------|
| Low Target | ~25-30 mg/dL (~2.2-2.7 mmo | l/L) ~10-15 mg/L |
| Medium Target | ~200 mg/dL (~18 mmol/L) | ~40 mg/L |
| High Target | ~ 400-450 mg/dL (~35-40 mmol/ | ′L) ~150-200 mg/L |

- 6. Ensure adequate mixing before analysis.
- 7. Cartridges are stored at 4° each cartridge requires 10-15 mins warm up time so consider this requirement when planning study needs.
- 8. Run each level in duplicate on the Allegro using the same channel to reduce variability
- 9. Collect, review and collate data
- 10. Total Analysis Time: 7 mins x 6 = 42 mins in morning, 7 mins x 6 = 42 mins in afternoon plus preparation time

#### Data Analysis

The between-day precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1, 2].

#### **Data Review**

This data will be summarized in a final report which will also include an assessment of the accuracy. This report should be reviewed by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of Allegro performance prior to the conductance of clinical studies.

## References

1. Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

# **Between-Day Precision Study Data Collection Sheet**

| Hospital Name: | Date of Study: |
|-------------------------|----------------------------------------|
| Reference Analyzer | |
| Level 1 Urine Creatinin | e and Urine Δlhumin |
| Morning | e and office Albamin |
| | sult: Urine Creatinine mg/dL or mmol/L |
| Reference Analyzer Res | sult: Urine Albumin mg/L or g/L |
| <u>Afternoon</u> | |
| Reference Analyzer Re | sult: Urine Creatinine mg/dL or mmol/L |
| Reference Analyzer Re | sult: Uring Albumin mg/L or g/L |

| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | |
| | Cartridge Lot # | | | | | | | | |
| Low QC | Range: | | | | | | | | |
| High QC | Range: | | | | | | | | |
| | | | Mor | ning | | | After | noon | |
| | | Urine Creat | Urine Creat | Urine | Urine | Urine Creat | Urine Creat | Urine | Urine |
| | | Result | Result | Albumin | Albumin | Result | Result | Albumin | Albumin |
| | | mg/dL or | mg/dL or | Result | Result | mg/dL or | mg/dL or | Result | Result |
| | Replicate # | mmol/L | mmol/L | mg/L or g/L | mg/L or g/L | mmol/L | mmol/L | mg/L or g/L | mg/L or g/L |
| | Day 1 | | | | | | | | |
| | Day 2 | | | | | | | | |
| | Day 3 | | | | | | | | |
| | Day 4 | | | | | | | | |
| | Day 5 | | | | | | | | |
| | Day 6 | | | | | | | | |
| | Day 7 | | | | | | | Ī | |
| | Day 8 | | | | | | | | |
| | Day 9 | | | | | | | | |
| | Day 10 | | | | | | | | |

# Level 2 Urine Creatinine and Urine Albumin

| <u>Morning</u> | |
|-------------------------------------------------------------|---|
| Reference Analyzer Result: Urine Creatinine mg/dL or mmol/L | |
| Reference Analyzer Result: Urine Albumin mg/L or g/L | _ |
| <u>Afternoon</u> | |
| Reference Analyzer Result: Urine Creatinine mg/dL or mmol/L | |
| Reference Analyzer Result: Urine Albumin mg/L or g/L | |

| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | |
| | Cartridge Lot # | | | | | | | | |
| Low QC | Range: | | | | | | | | |
| High QC | Range: | | | | | | | | |
| | | | Mor | ning | | | After | noon | |
| | Replicate # | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine<br>Albumin<br>Result<br>mg/L or g/L |
| | Day 1 | | | <u> </u> | <u> </u> | | | <u> </u> | G. G. |
| | Day 2 | | | | | | | | |
| | Day 3 | | | | | | | | |
| | Day 4 | | | | | | | | |
| | Day 5 | | | | | | | | |
| | Day 6 | | | | | | | | |
| | Day 7 | | | | | | | | |
| | Day 8 | | | | | | | | |
| | Day 9 | | | | | | | | |
| | Day 10 | | | | | | | | |

| Morning | | | | |
|---|---|---|---|---|
| Reference Ar | nalyzer Result: Ur | ine Creatinin | e mg/dL or m | nmol/L |
| Reference Ar | nalyzer Result: Ur | ine Albumin | mg/L or g/L | |
| <u>Afternoon</u> | | | | |
| Reference Ar | nalyzer Result: Ur | ine Creatinin | e mg/dL or m | nmol/L |
| Reference Ar | nalyzer Result: Ur | ine Albumin | mg/L or g/L | |
| | System Name | | | |
| | System Serial # | | | |

| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | |
| | Cartridge Lot # | | | | | | | | |
| Low QC | Range: | | | | | | | | |
| High QC | Range: | | | | | | | | |
| | | | | ning | | | After | noon | |
| | Replicate # | Urine Creat<br>Result | Urine Creat<br>Result | Urine<br>Albumin | Urine<br>Albumin | Urine Creat<br>Result | Urine Creat<br>Result | Urine<br>Albumin | Urine<br>Albumin |
| | | mg/dL or | mg/dL or | Result | Result | mg/dL or | mg/dL or | Result | Result |
| | | mmol/L | mmol/L | mg/L or g/L | mg/L or gl/L | mmol/L | mmol/L | mg/L or gl/L | mg/L or g/L |
| | Day 1 | | | | | | | | |
| | Day 2 | | | | | | | | |
| | Day 3 | | | | | | | | |
| | Day 4 | | | | | | | | |
| | Day 5 | | | | | | | | |
| | Day 6 | | | | | | | | |
| | Day 7 | | | | | | | | |
| | Day 8 | | | | | | | | |
| | Day 9 | | | | | | | | |
| | Day 10 | | | | | | | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |

| I. Urine Creatinine and Urine Albumin | |
|---|---|
| III. Method Comparison Study Protocol | |
| Protocol based on the following guidance documents: | |
| Clinical & Laboratory Standards Institute (CLSI). Method Comparison and Bias Estimation Using Patient Sam<br>Approved Guideline – Second Edition. EP9-A2. | ıples |

# **Purpose**

This protocol is designed to investigate how Allegro results compare to a recognized central laboratory reference method. These studies are important in order to establish the relationship between the Allegro System and the reference method with respect to statistical correlation and measurement bias. This protocol is designed and recommended for the Allegro System.

# **Background**

Good practice dictates that the performance of medical devices such as the Allegro System be verified before the conductance of clinical studies. Verification studies include: method comparisons to determine how the results of the Allegro Systems compare to a recognized reference method, studies of imprecision to determine the reproducibility of the various tests available on the Allegro, and to determine the analytical trueness of the Allegro measurements. The protocol below describes how to conduct a method comparison (Allegro vs. Reference Method).

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Kidney Function Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic tubes for decanting urine samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

**Tests:** Urine Creatinine and urine Albumin

Sample Type: Fresh random urine

Sample Size: 25μL Time per UABCR: 7 mins

**Linear Range of Operation:** 15-500 mg/dL (13.0-44.2 mmol/L) **Linear Range of Operation for Urine Albumin:** 3-300 mg/L

#### **Expected Normal Values**

Urine Creatinine: For a random urine sample, >12 Years Male 20-370 mg/dL (1.8- 32.7 mmol/L), >12 Years

Female 20 – 320 mg/dL (1.8-28.3 mmol/L)

Urine Albumin: For a random urine sample, normal values are typically 0 to 30 mg/L

# **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

**Urine Albumin and Creatinine:** 

Low Level Target: Urine Albumin ~50 mg/L Creatinine ~85mg/dL (~8 mmol/L)

High Level Target: Urine Albumin ~180 mg/L Creatinine ~220 mg/dL (~20 mmol/L)

Please note that urine creatinine and urine Albumin are processed at the same time and can be run in both channels

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. 40-50 fresh (within 24hrs) discarded random urine samples should be collected and run in duplicate on Allegro. Again spiking with creatinine spiking solutions and human Albumin may be required to cover the measuring range.
- 4. Ensure adequate mixing before analysis.
- 5. Samples should be analysed promptly on the reference analyser.
- 7. Cartridges are stored at 4° each cartridge requires 10-15 mins warm up time so consider this requirement when planning study needs.
- 8. Analyse all samples in duplicate on the Allegro using the same channel to reduce variability
- 9. Collect, Review and collate data.
- 10. Total Analysis Time: 7 mins x 80-100 = 560 700 mins. Approx. 9.3 11.6 hrs plus preparation time
- 11. To reduce analysis time consider running samples in singles or perhaps less samples in duplicate whichever best suits site

#### **Data Analysis**

As part of this study paired urine creatinine and urine Albumin measurements will be collected. Analysis of accuracy is based on pairing individual results from the Allegro with the corresponding reference analyser measurement and calculating the difference (bias). Scatter plots and linear regression analysis are appropriate tools to assess the relationship between the Allegro results and the reference analyzer. Moreover Bland-Altman plots can be used to assess the bias relative to the range of urine creatinine and urine Albumin concentrations studied. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1, 2]. The validity of the conclusions is dependent on experimental design, chiefly number of samples, the distribution of results, and the calibration of the reference analyzer.

#### **Data Review**

This data will be summarized in a summary report which will also include an assessment of precision. This report should be reviewed and signed off by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of the Allegro System performance prior to the conductance of clinical studies.

#### References

1. Clinical & Laboratory Standards Institute (CLSI). *Method Comparison and Bias Estimation Using Patient Samples; Approved Guideline – Second Edition. EP9-A2.* 

| Study Site: | Date of Study: |
|-----------------------|----------------|
| System Operator(s): | |
| Specimen Type (Urine) | |
| Reference Analyzer | |

| | 1 | | ı | ı | ı | ı |
|---|---|---|---|---|---|---|
| | System Name | | | | | |
| | System Serial # | | | | | |
| | Cartridge Lot # | | | | | |
| Low QC | Range: | | | | | |
| High QC | Range: | | | | | |
| Specimen ID | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Urine<br>Creat mg/dL<br>or mmol/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Reference<br>Analyser<br>Result Urine<br>Albumin mg/L<br>or g/L |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| 5 | | | | | | |
| 6 | | | | | | |
| 7 | | | | | | |
| 8 | | | | | | |
| 9 | | | | | | |
| 10 | | | | | | |
| 11 | | | | | | |
| 12 | | | | | | |
| 13 | | | | | | |
| 14 | | | | | | |
| 15 | | | | | | |
| 16 | | | | | | |
| 17 | | | | | | |
| 18 | | | | | | |
| 19 | | | | | | |
| 20 | | | | | | |
| 21 | | | | | | |
| 22 | | | | | | |
| 23 | | | | | | |
| 24 | | | | | | |
| 25 | | | | | | |
| 26 | | | | | | |

| 27 |
|----|
| 28 |
| 29 |
| 30 |

# **Method Comparison Data Collection Sheet (Case Report Form)**


| | | | I | I | | - |
|---|---|---|---|---|---|---|
| | System Name | | | | | |
| | System Serial # | | | | | |
| | Cart Lot # | | | | | |
| Specimen ID | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Urine<br>Creat mg/dL<br>or mmol/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Reference<br>Analyser<br>Result Urine<br>Albumin mg/L<br>or g/L |
| 31 | | | | | | |
| 32 | | | | | | |
| 33 | | | | | | |
| 34 | | | | | | |
| 35 | | | | | | |
| 36 | | | | | | |
| 37 | | | | | | |
| 38 | | | | | | |
| 39 | | | | | | |
| 40 | | | | | | |
| 41 | | | | | | |
| 42 | | | | | | |
| 43 | | | | | | |
| 44 | | | | | | |
| 45 | | | | | | |
| 46 | | | | | | |
| 47 | | | | | | |
| 48 | | | | | | |
| 48 | | | | | | |
| 49 | | | | | | |
| 50 | | | | | | |
| 51 | | | | | | |
| 52 | | | | | | |
| 53 | | | | | | |
| 54 | | | | | | |
| 55 | | | | | | |
| 56 | | | | | | |
| 57 | | | | | | |
| 58 | | | | | | |
| 59 | | | | | | |
| 60 | | | | | | |
| 61 | | | | | | |
| 62 | | | | | | |
| 63 | | | | | | |
| 64 | | | | | | |
| 65 | | | | | | |

| 66 |
|----|
| 67 |
| 68 |
| 69 |
| 70 |
| 71 |
| 72 |

Method Comparison Data Collection Sheet (Case Report Form)


| | System Name | | | | | |
|---|---|---|---|---|---|---|
| | System Serial | | | | | |
| | # | | | | | |
| | Cart Lot # | | | | | |
| Specimen ID | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Urine Creat<br>Result<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Urine<br>Creat mg/dL<br>or mmol/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Urine<br>Albumin<br>Result<br>mg/L or g/L | Reference<br>Analyser<br>Result Urine<br>Albumin mg/L<br>or g/L |
| 73 | | | | | | |
| 74 | | | | | | |
| 75 | | | | | | |
| 76 | | | | | | |
| 77 | | | | | | |
| 78 | | | | | | |
| 79 | | | | | | |
| 80 | | | | | | |
| 81 | | | | | | |
| 82 | | | | | | |
| 83 | | | | | | |
| 84 | | | | | | |
| 85 | | | | | | |
| 86 | | | | | | |
| 87 | | | | | | |
| 88 | | | | | | |
| 89 | | | | | | |
| 90 | | | | | | |
| 91 | | | | | | |
| 92 | | | | | | |
| 93 | | | | | | |
| 94 | | | | | | |
| 95 | | | | | | |
| 96 | | | | | | |
| 97 | | | | | | |
| 98 | | | | | | |
| 99 | | | | | | |
| 100 | | | | | | |

# 1. Urine Creatinine and Urine Albumin Summary Report Template

| rine Creatinine and Urine Albumin Summary Report |
|--------------------------------------------------|
| Date: |
| Report Author: |
| Study Site: |
| Study Site Principal Investigator/Department: |

# **Materials and Methods**

See Protocols I-IV. Any deviations from protocol should be noted here.

# **Summary of Results**

# I. Precision Studies

Table 1. Urine Creatinine Within-Day Precision for Allegro

| | Low Urine<br>Creat | Mid Urine<br>Creat | High Urine<br>Creat |
|---|---|---|---|
| Mean mg/dL or mmol/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix: Urine | | | |

Table 2. Urine Albumin Within-Day Precision for Allegro

| | Low Urine<br>Urine<br>Albumin | Mid Urine<br>Urine<br>Albumin | High Urine<br>Urine<br>Albumin |
|---|---|---|---|
| Mean mg/L or g/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix: Urine | | | |

Table 3. Urine Creatinine Between-Day Precision for Allegro

| | Low Urine<br>Creat | Mid Urine<br>Creat | High Urine<br>Creat |
|---|---|---|---|
| Mean mg/dL or mmol/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix: Urine | | | |

Table 4. Urine Albumin Between-Day Precision for Allegro

| | Low Urine<br>Urine<br>Albumin | Mid Urine<br>Urine<br>Albumin | High Urine<br>Urine<br>Albumin |
|---|---|---|---|
| Mean mg/L or g/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix: Urine | | | |

# **II.** Method Comparison

Table 7. Summary of Linear Regression Analysis Results Urine creatinine and Urine Albumin for the Allegro

| | <b>Urine Creat</b> | <b>Urine Albumin</b> |
|---|---|---|
| Slope | | |
| y-intercept (mg/dL) | | |
| R <sup>2</sup> | | |
| N | | |
| Urine Creat Range mg/dL or mmol/L | | |
| Urine Albumin Range mg/L or g/L | | |

Table 8. Summary of Bland-Altman Results

| Mean Bias (mg/dL) |
|-----------------------------------|
| 95% Limits of Agreement |
| Lower |
| Upper |
| Urine Creat Range mg/dL or mmol/L |
| Urine Albumin Range mg/L or gl/L |

| Summary Findings | |
|------------------------------------------------|------|
| Allegro demonstrated | |
| This report has been reviewed and approved by: | |
| Signature of Study Site Principal Investigator | Date |
| Signature of MASA Director | Date |

# 2. HbA1c

I. Within Day Precision Study Protocol

Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

## **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the within-day precision of whole blood HbA1c measurements on the Allegro system.

# **Materials Needed**

- Nova Biomedical Allegro
- Allegro Glycaemic Control Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting EDTA samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips

Appropriate Spiking stock solutions

# **Important Factors to Consider**

Tests: HbA1c Sample Type:

- Capillary blood (from finger stick)
- Fresh venous whole blood with anticoagulants ethylenediamine tetra-acetic acid (EDTA); Li heparin; Na heparin

**Sample Size:** 1.5 μL

Time per HbA1c: 6.5 mins

Linear Range of Operation for HbA1c: 4-15% (20.2 - 140.4 mmol/L)

#### **Potential Interferences**

HbA1c measurement is not affected by Hb variants: HbAc, HbAD, HbAE, HbF, HbAG and HbAS

#### **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

HbA1c:

Low Level Target: ~5% (31.1 mmol/mol)

High Level Target: ~10% (85.5 mmol/mol)

**Normal Values** 

HbA1c: - A normal non-diabetic HbA1c is <5.5% (36mmol/mol). In diabetes about 6.5% (48 mmol/mol) is good.

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. Using aliquoted venous EDTA whole blood identify three levels low, medium and high.
- 4. Suggested concentrations for low, medium and high samples: -

HbA1c

Low Target ~5% (31.1 mmol/mol) Medium Target ~7% (53 mmol/mol)

32

Version 3: 18 July 2016

- 5. Ensure adequate mixing before analysis.
- 6. Cartridges are stored at 4° each cartridge the HbA1c cartridge can be used cold
- 7. Run each Level <u>10</u> times on Allegro, the HbA1c cartridge can only be run in the 600nm channel which is on the right hand side of the analyser.
- 8. Collect, review and collate data.

**Total Analysis Time:** 6.25 mins x 10 = 62.5 mins per level. 187.5 mins for all levels. Approx. 3.15 hrs plus preparation time

# **Data Analysis**

The within-run precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [4].

#### **Data Review**

This data will be summarized in a final report which will also include an assessment of the accuracy. This report should be reviewed by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of Allegro performance prior to the conductance of clinical studies.

#### References

1. Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

# Appendix 1

# 

| | % or mmol/Mol |
|----|---------------|
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | |
| 9 | |
| 10 | |

# Level 2 HbA1c

Reference Analyzer Result % or mmol/mol \_\_\_\_\_

| | System Name | |
|---------|-----------------|------------------------|
| | System Serial # | |
| | Cartridge Lot # | |
| Low QC | Range: | |
| High QC | Range: | |
| | Replicate # | HbA1c<br>% or mmol/mol |
| | 1 | |
| | 2 | |
| | 3 | |
| | 4 | |
| | 5 | |
| | 6 | |
| | 7 | |
| | 8 | |

| 9 |
|----|
| 10 |

# Level 3 HbA1c

Reference Analyzer Result % or mmol/mol\_\_\_\_\_

| | System Name | |
|---------|-----------------|------------------------|
| | System Serial # | |
| | Cartridge Lot # | |
| Low QC | Range: | |
| High QC | Range: | |
| | Replicate # | HbA1c<br>% or mmol/mol |
| | 1 | |
| | 2 | |
| | 3 | |
| | 4 | |
| | 5 | |
| | 6 | |
| | 7 | |
| | 8 | |
| | 9 | |
| | 10 | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |
## 2. HbA1c

### II. Between-Day Precision Study Protocol

#### Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). *Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition.* EP5-A2.

#### **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the between-day precision of whole blood HbA1c measurements on the Allegro system.

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Glycemic Control Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting EDTA samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips

If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

## Tests: HbA1c Sample Type:

- Capillary blood (from finger stick)
- Fresh venous whole blood with anticoagulants ethylenediamine tetra-acetic acid (EDTA); Li heparin; Na heparin

Sample Size: 1.5 µL

Time per HbA1c: 6.5 mins

Linear Range of Operation for HbA1c: 4-15% (20.2 - 140.4 mmol/L)

#### **Potential Interferences**

HbA1c measurement is not affected by Hb variants: HbAc, HbAD, HbAE, HbF, HbAG and HbAS

#### **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

#### HbA1c:

Low Level Target: ~5% (~31.1 mmol/mol)

High Level Target: ~10% (~85.8 mmol/mol)

#### **Normal Values**

HbA1c:- A normal non-diabetic HbA1c is <5.5% (36mmol/mol). In diabetes about 6.5% (48 mmol/mol) is good.

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Analyse controls on Allegro every day that testing is carried out, 2 runs per day would be performed one in the morning and the other in the afternoon so QC would need to be performed prior to each run, make sure results are within specification before proceeding. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.

- 3. Because of the logistical difficulty of using whole blood over a 2-week period the suggestion here is to use the Control Solutions, these provide only 2 levels, but these should be aliquoted into  $40 \times 50 \mu L$  aliquots and frozen to reduce variables.
- 4. A freshly aliquot will be thawed, mixed and analysed every morning and afternoon in duplicate for 10 consecutive working days.
- 6. Cartridges are stored at 4° each cartridge the HbA1c cartridge can be used cold
- 7. Run each Level in duplicate on Allegro, the HbA1c cartridge can only be run in the 600nm channel which is on the right hand side of the analyser.
- 8. Collect, review and collate data

**Total Analysis Time:** 6.25 mins x 4 = 25 mins in morning, 6.25 mins x 4 = 25 mins in afternoon. Approx. 50 mins plus preparation time

#### **Data Analysis**

The between-day precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1].

#### **Data Review**

This data will be summarized in a final report which will also include an assessment of the accuracy. This report should be reviewed by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of Allegro performance prior to the conductance of clinical studies.

#### References

1. Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

#### Appendix 2

#### **Between-Day Precision Study Data Collection Sheet**

| Hospital Name:System Operator(s): | Date of Study: |
|-----------------------------------------------------------|----------------|
| Reference Analyzer | |
| Level 1 HbA1c | |
| Morning Reference Analyzer Result % or mmol/mol Afternoon | |

| | System Name | | | | |
|---|---|---|---|---|---|
| | System Serial # | | | | |
| | Cartridge Lot # | | | | |
| Low QC | Range: | | | | |
| High QC | Range: | | | | |
| | | Mor | ning | After | noon |
| | Replicate # | HbA1c Result<br>% or<br>mmol/mol | HbA1c Result<br>% or<br>mmol/mol | HbA1c Result<br>% or<br>mmol/mol | HbA1c Result<br>% or<br>mmol/mol |
| | Day 1 | | | | |
| | Day 2 | | | | |
| | Day 3 | | | | |
| | Day 4 | | | | |
| | Day 5 | | | | |
| | Day 6 | | | | |
| | Day 7 | | | | |
| | Day 8 | | | | |
| | Day 9 | | | | |
| | Day 10 | | | | |

#### Level 2 HbA1c

| Morning |
|-----------------------------------------|
| Reference Analyzer Result % or mmol/mol |
| <u>Afternoon</u> |
| Reference Analyzer Result % or mmol/mol |

| | System Name | | | | |
|---------|-----------------|-----|------|-------|------|
| | System Serial # | | | | |
| | Cartridge Lot # | | | | |
| Low QC | Range: | | | | |
| High QC | Range: | | | | |
| | | Mor | ning | After | noon |

| | HbA1c Result | HbA1c Result | HbA1c Result | HbA1c Result |
|-------------|--------------|--------------|--------------|--------------|
| Replicate # | % or | % or | % or | % or |
| | mmol/mol | mmol/mol | mmol/mol | mmol/mol |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Day 4 | | | | |
| Day 5 | | | | |
| Day 6 | | | | |
| Day 7 | | | | |
| Day 8 | | | | |
| Day 9 | | | | |
| Day 10 | | | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |

| | | ١. | | 4 | |
|---|---|----|---|---|---|
| , | Н | n | Λ | 1 | r |
| | | u | _ | | |

III. Method Comparison Study Protocol

Protocol based on the following guidance documents:

Clinical & Laboratory Standards Institute (CLSI). *Method Comparison and Bias Estimation Using Patient Samples;*Approved Guideline – Second Edition. EP9-A2.

#### **Purpose**

This protocol is designed to investigate how Allegro results compare to a recognized central laboratory reference method. These studies are important in order to establish the relationship between the Allegro System and the reference method with respect to statistical correlation and measurement bias. This protocol is designed and recommended for the Allegro System.

#### **Background**

Good practice dictates that the performance of medical devices such as the Allegro System be verified before the conductance of clinical studies. Verification studies include: method comparisons to determine how the results of the Allegro Systems compare to a recognized reference method, studies of imprecision to determine the reproducibility of the various tests available on the Allegro to determine the analytical trueness of the Allegro measurements. The protocol below describes how to conduct a method comparison (Allegro vs. Reference Analyser).

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Glycaemic Control Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting EDTA samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

Tests: HbA1c Sample Type:

Capillary blood (from finger stick)

 Fresh venous whole blood with anticoagulants ethylenediamine tetra-acetic acid (EDTA); Li heparin; Na heparin

Sample Size: 1.5 µL

Time per HbA1c: 6.25 mins

Linear Range of Operation for HbA1c: 4-15% (20.2 - 140.4 mmol/L)

#### **Potential Interferences**

HbA1c measurement is not affected by Hb variants: HbAc, HbAD, HbAE, HbF, HbAG and HbAS

#### **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

#### HbA1c:

Low Level Target: ~5% (~31.1 mmol/mol)

High Level Target: ~10% (~85.5 mmol/mol)

#### **Normal Values**

HbA1c:- A normal non-diabetic HbA1c is <5.5% (36mmol/mol). In diabetes about 6.5% (48 mmol/mol) is good.

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. Select 40-50 fresh discarded HbA1c EDTA samples that cover the measuring range if possible.
- 4. Ensure adequate mixing before analysis.
- Cartridges are stored at 4° each cartridge the HbA1c cartridge can be used cold
- 6. Run all samples in duplicate on Allegro following analysis on the reference analyser. Cartridges Allegro, the HbA1c cartridge can only be run in the 600nm channel which is on the right hand side of the analyser.
- 7. Collect, Review and collate data.
- 8. Total Analysis Time:  $6.25 \text{ mins } \times 80 100 = 500 625 \text{ mins.}$  Approx. 8.3 10.4 hrs plus preparation time
- 9. To reduce analysis time consider running samples in singles or perhaps less samples in duplicate whichever best suits site

#### **Data Analysis**

As part of this study paired HbA1c measurements will be collected. Analysis of accuracy is based on pairing individual results from the Allegro with the corresponding reference analyser measurement and calculating the difference (bias). Scatter plots and linear regression analysis are appropriate tools to assess the relationship between the Allegro results and the reference analyzer. Moreover, Bland-Altman plots can be used to assess the bias relative to the range studied. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [2]. The validity of the conclusions is dependent on experimental design, chiefly number of samples, the distribution of results, and the calibration of the reference analyzer.

#### **Data Review**

This data will be summarized in a summary report which will also include an assessment of precision. This report should be reviewed and signed off by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of the Allegro System performance prior to the conductance of clinical studies.

#### References

1. Clinical & Laboratory Standards Institute (CLSI). Method Comparison and Bias Estimation Using Patient Samples; Approved Guideline – Second Edition. EP9-A2.

## **Method Comparison Data Collection Sheet (Case Report Form)**

| Study Site: | Date of Study: |
|-----------------------------------------|----------------|
| System Operator(s): | |
| Specimen Type (Venous EDTA Whole Blood) | |
| Reference Analyzer | |

| | System Name | | |
|-----------------|-------------------|--------------|--------------|
| System Serial # | | | |
| | Cartridge Lot # | | |
| Low QC | Range: | | |
| High QC | Range: | | |
| | Reference | HbA1c result | HbA1c result |
| Specimen ID | Analyzer Result % | % or | % or |
| | or mmol/mol | mmol/mol | mmol/mol |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| 5 | | | |
| 6 | | | |
| 7 | | | |
| 8 | | | |
| 9 | | | |
| 10 | | | |
| 11 | | | |
| 12 | | | |
| 13 | | | |
| 14 | | | |
| 15 | | | |
| 16 | | | |
| 17 | | | |
| 18 | | | |
| 19 | | | |
| 20 | | | |
| 21 | | | |
| 22 | | | |
| 23 | | | |
| 24 | | | |
| 25 | | | |
| 26 | | | |
| 27 | | | |
| 28 | | | |
| 29 | | | |
| 30 | | | |

| | 1 | | · |
|---|---|---|---|
| | System Name | | |
| | System Serial # | | |
| | Cart Lot # | | |
| | Reference | HbA1c result | HbA1c result |
| Specimen ID | Analyzer Result % or mmol/mol | % or<br>mmol/mol | % or<br>mmol/mol |
| 31 | | • | -, - |
| 32 | | | |
| 33 | | | |
| 34 | | | |
| 35 | | | |
| 36 | | | |
| 37 | | | |
| 38 | | | |
| 39 | | | |
| 40 | | | |
| 41 | | | |
| 42 | | | |
| 43 | | | |
| 44 | | | |
| 45 | | | |
| 46 | | | |
| 47 | | | |
| 48 | | | |
| 48 | | | |
| 49 | | | |
| 50 | | | |
| 51 | | | |
| 52 | | | |
| 53 | | | |
| 54 | | | |
| 55 | | | |
| 56 | | | |
| 57 | | | |
| 58 | | | |
| 59 | | | |
| 60 | | | |
| 61 | | | |
| 62 | | | |
| 63 | | | |
| 64 | | | |
| 65 | | | |
| 66<br>67 | | | |
| 68 | | | |
| 69 | | | |
| 70 | | | |
| 70 | | | |
| 72 | | | |
| 73 | | | |
| /3 | | | |

| | 1 | | 1 |
|---|---|---|---|
| | System Name | | |
| | System Serial # | | |
| | Cart Lot # | | |
| Specimen ID | Reference<br>Analyzer Result %<br>or mmol/mol | HbA1c result<br>% or<br>mmol/mol | HbA1c result<br>% or<br>mmol/mol |
| 74 | | - | |
| 75 | | | |
| 76 | | | |
| 77 | | | |
| 78 | | | |
| 79 | | | |
| 80 | | | |
| 81 | | | |
| 82 | | | |
| 83 | | | |
| 84 | | | |
| 85 | | | |
| 86 | | | |
| 87 | | | |
| 88 | | | |
| 89 | | | |
| 90 | | | |
| 91 | | | |
| 92 | | | |
| 93 | | | |
| 94 | | | |
| 95 | | | |
| 96 | | | |
| 97 | | | |
| 98 | | | |
| 99 | | | |
| 100 | | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |

# 2. HbA1c Summary Report Template

| Date: |
|-----------------------------------------------|
| Report Author: |
| Study Site: |
| Study Site Principal Investigator/Department: |

**Materials and Methods** 

**HbA1c Summary Report** 

See Protocols I-IV. Any deviations from protocol should be noted here.

## **Summary of Results**

#### I. Precision Studies

Table 1. **HbA1c Within-Day** Precision for Allegro

| | Low HbA1c | Mid HbA1c | High HbA1c |
|--------------------|-----------|-----------|------------|
| Mean % or mol/mol | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 2. HbA1c Between-Day Precision for Allegro

| | Low HbA1c | Mid HbA1c | High HbA1c |
|--------------------|-----------|-----------|------------|
| Mean % or mol/mol | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

## **II.** Method Comparison

Table 5. Summary of Linear Regression Analysis Results HbA1C for Allegro

| | HbA1c |
|------------------------------|-------|
| Slope | |
| y-intercept (% or mmol/mol)) | |
| R <sup>2</sup> | |
| N | |
| HbA1c Range % or mmol/mol | |

Table 6. Summary of Bland-Altman Results

| | HbA1c |
|---------------------------|-------|
| Mean Bias (% or mmol/mol) | |
| 95% Limits of Agreement | |
| Lower | |
| Upper | |
| HbA1c (% or mmol/mol) | |

## **Summary Findings**

Allegro demonstrated ....

This report has been reviewed and approved by:

| Signature of Study Site Principal Investigator | Date |
|--------------------------------------------------|--------|
| Signature of MASA Director | Date |
| 3. Total Cholesterol, Triglyceride and HDL Chole | sterol |

Within Day Precision Study Protocol ١.

Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition. EP5-A2.

#### **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the within day precision of whole blood total cholesterol, triglycerides and HDL cholesterol measurements on the Allegro system.

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Lipid Risk Cartridges
- Nova Biomedical Allegro Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting Na Heparin or Li Heparin samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

**Tests:** Total Cholesterol, Triglycerides, HDL Cholesterol

Sample Type: Subject to change but to date:

- Capillary whole blood (from finger stick)
- Venous whole blood with anticoagulants Na heparin; Li heparin
- Venous plasma with anticoagulants Na heparin; Li heparin

Serum

Sample Size: 5 µL

Time per Lipid: 10 mins

Linear Range of Operation for Total Cholesterol: 100-450 mg/dL (2.59-11.64 mmol/L)

Linear Range of Operation for Triglyceride: 50-600 mg/dL (0.56-6.76 mmol/L)

Linear Range of Operation for HDL Cholesterol: 20-100 mg/dL (0.52- 2.59 mmol/L)

Please note that all parameters are processed at the same time.

#### **Normal Values:**

**Total Cholesterol:** Desirable is below 200 mg/dL (<5.17 mmol/L) **Triglycerides:** Desirable is below 150 mg/dL (<1.69 mmol/L) **HDL Cholesterol:** Desirable is 60 mg/dL and above (> 1.55 mg/dL)

## **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

| | <b>Total Cholesterol</b> | Triglycerides | HDL Cholesterol |
|---|---|---|---|
| Low Level Target: | ~ 170 mg/dL | ~150 mg/dL | ~40 mg/dL |
| | (~4.40 mmol/L) | (~1.69 mmol/L) | (~1.04 mmol/L) |
| High Level Target: | ~ 240 mg/dL | ~300 mg/dL | ~60 mg/dL (1.55 mmol/L) |
| | (~6.21 mmol/L) | (~3.39 mmol/L) | (~1.55 mmol/L) |

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. If possible using fresh aliquoted venous Na or Lithium heparin whole blood samples from qualified patients identify levels low, medium and high Total Cholesterol, Triglycerides and HDL Cholesterol levels.
- 4. Suggested concentrations for low, medium and high samples: -

| | <b>Total Cholesterol</b> | Triglycerides | <b>HDL Cholesterol</b> |
|---|---|---|---|
| Low Level Target: | ~ 150 mg/dL | ~100 mg/dL | ~40 mg/dL |
| | (~3.88 mmol/L) | (~1.13mmol/L) | (~1.03 mmol/L) |
| Medium Level Target: | ~ 250 mg/dL | ~200 mg/dL | ~60 mg/dL |
| | (~6.47 mmol/L) | (~2.26 mmol/L) | (~1.55 mmol/L) |
| High Level Target: | ~ 400 mg/dL | ~300 mg/dL | ~80 mg/dL |
| | (~10.35 mmol/L) | ~3.39 mmol/L) | (~2.07 mmol/L) |

- Cartridges are stored at 4° each cartridge the HbA1c cartridge can be used cold
- 3. Cartridges are stored at 4° each cartridge the lipids cartridge is only stable at RT for 1 hour
- 4. Run each Level <u>10</u> times on Allegro, the Lipids cartridge can only be run in the 660nm channel which is on the left hand side of the analyser.
  - 6. Collect, review and collate data

**Total Analysis time:** 10 x 10 mins=100 mins per level. 300 mins for all levels this is just run time. Approx. 5 hrs. plus preparation time

#### **Data Analysis**

The within-run precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1, 2].

#### **Data Review**



Appendix 1

Within-Day Precision Study Data Collection Sheet

| Hospital Name: | Date of Study: |
|------------------------------------------|-------------------------|
| System Operator(s): | |
| Reference Analyzer | <del></del> |
| Level 1 Total Cholesterol, Triglycerides | and HDL Cholesterol |
| Reference Analyzer Result mg/dL or m | mol/L Total Cholesterol |
| Reference Analyzer Result mg/dL or m | mol/L Triglycerides |
| Reference Analyzer Result mg/dL or m | mol/L HDL Cholesterol |

| | System Name | | | |
|---|---|---|---|---|
| | System Serial # | | | |
| | Cartridge Lot # | | | |
| Low QC | Range: | | | |
| High QC | Range: | | | |
| | Replicate # | Total<br>Cholesterol<br>mg/dL or<br>mmol/L | Triglycerides<br>mg/dL or<br>mmol/L | HDL Cholesterol<br>mg/dL or<br>mmol/L |
| | 1 | | | |
| | 2 | | | |
| | 3 | | | |
| | 4 | | | |
| | 5 | | | |
| | 6 | | | |
| | 7 | | | |
| | 8 | | | |
| | 9 | | | |
| | 10 | | | |

#### <u>Level 2 Total Cholesterol, Triglycerides and HDL Cholesterol</u>

Reference Analyzer Result mg/dL or mmol/L Total Cholesterol \_\_\_\_\_\_ Reference Analyzer Result mg/dL or mmol/L Triglycerides \_\_\_\_\_

| Reference Analyzer Result mg/dL or mmol/L HDL Cholesterol |
|-----------------------------------------------------------|
|-----------------------------------------------------------|

| | System Name | | | |
|---|---|---|---|---|
| | System Serial # | | | |
| | Cartridge Lot # | | | |
| Low QC | Range: | | | |
| High QC | Range: | | | |
| | Replicate # | Total<br>Cholesterol<br>mg/dL or<br>mmol/L | Triglycerides<br>mg/dL or<br>mmol/L | HDL Cholesterol<br>mg/dL or<br>mmol/L |
| | 1 | | | |
| | 2 | | | |
| | 3 | | | |
| | 4 | | | |
| | 5 | | | |
| | 6 | | | |
| | 7 | | | |
| | 8 | | | |
| | 9 | | | |
| | 10 | | | |

## Level 3 Total Cholesterol, Triglycerides and HDL Cholesterol

| Reference Analyzer Result mg/dL or mmol/L Total Cholesterol _ |
|---------------------------------------------------------------|
| Reference Analyzer Result mg/dL or mmol/L Triglycerides |
| Reference Analyzer Result mg/dL or mmol/L HDL Cholesterol |

| | System Name | | | |
|---|---|---|---|---|
| | System Serial # | | | |
| | Cart Lot # | | | |
| Low QC | Range: | | | |
| High QC | Range: | | | |
| | Replicate # | Total<br>Cholesterol<br>mg/dL or<br>mmol/L | Triglycerides<br>mg/dL or<br>mmol/L | HDL Cholesterol<br>mg/dL or<br>mmol/L |
| | 1 | | | |
| | 2 | | | |
| | 3 | | | |
| | 4 | | | |
| | 5 | | | |
| | 6 | | | |
| | 7 | | | |
| | 8 | | | |
| | 9 | | | |
| | 10 | | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Data: |

| 3. Total Cholesterol, Triglyceride and HDL Choles | stero |
|---------------------------------------------------|-------|
|---------------------------------------------------|-------|

II. Between-Day Precision Study Protocol

Protocol based on:

Clinical & Laboratory Standards Institute (CLSI). *Evaluation of Precision Performance of Quantitative Measurement Methods; Approved Guideline – Second Edition.* EP5-A2.

#### **Purpose**

This protocol is recommended and designed by Nova Biomedical to investigate the between-day precision of urine creatinine and urine albumin measurements on the Allegro system.

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Lipid Cartridges
- Nova Biomedical Allegro Lipid Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting Na Heparin or Li Heparin samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

**Tests:** Total Cholesterol, Triglycerides, HDL Cholesterol

Sample Type: Subject to change but to date:

- Capillary whole blood (from finger stick)
- Venous whole blood with anticoagulants Na heparin; Li heparin
- Venous plasma with anticoagulants Na heparin; Li heparin

Serum

Sample Size: 5 µL

Time per Lipid: 10 mins

Linear Range of Operation for Total Cholesterol: 100-450 mg/dL (2.59-11.64 mmol/L)

**Linear Range of Operation for Triglyceride:** 50-600 mg/dL (0.56-6.76 mmol/L) **Linear Range of Operation for HDL Cholesterol:** 20-100 mg/dL (0.52- 2.59 mmol/L)

Please note that all parameters are processed at the same time.

#### **Normal Values:**

**Total Cholesterol:** Desirable is below 200 mg/dL (<5.17 mmol/L) **Triglycerides:** Desirable is below 150 mg/dL (<1.69 mmol/L) **HDL Cholesterol:** Desirable is 60 mg/dL and above (> 1.55 mg/dL)

#### **Accuracy Expectations**

**Total Cholesterol:** Target value  $\pm$  3% Triglycerides: Target value  $\pm$  5% **HDL Cholesterol:** Target value  $\pm$  5%

## **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

| | <b>Total Cholesterol</b> | Triglycerides | HDL Cholesterol |
|---|---|---|---|
| Low Level Target: | ~ 170 mg/dL | ~150 mg/dL | ~40 mg/dL |
| | (~4.40 mmol/L) | (~1.69 mmol/L) | (~1.04 mmol/L) |
| High Level Target: | ~ 240mg/dL | ~300 mg/dL | ~60 mg/dL (1.55 mmol/L) |
| | (~6.21 mmol/L) | (~3.39 mmol/L) | (~1.55 mmol/L) |

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- 2. Perform quality control runs on the Allegro being evaluated and the reference analyzer. Analyse controls on Allegro every day that testing is carried out, 2 runs per day would be performed one in the morning and the other in the afternoon so QC would need to be performed prior to each run, make sure results are within specification before proceeding. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. Because of the logistical difficulty of using whole blood over a 2-week period the suggestion here is to use the Control Solutions, these provide only 2 levels, but these should be aliquoted into  $40 \times 50 \mu L$  aliquots and frozen to reduce variables.

Note: If Allegro can analyse plasma then the samples used for within day precision can be centrifuged, aliquoted into 40 x 50µL microcentrifuge tubes, and frozen.

- 4. A freshly thawed aliquot will then be analysed every morning and afternoon in duplicate for 10 consecutive working days
- 5. Ensure adequate mixing before analysis.
- 5. Cartridges are stored at 4° each cartridge the lipids cartridge is only stable at RT for 1 hour
- 6. Run each Level in duplicate on the Allegro, the Lipids cartridge can only be run in the 660nm channel which is on the left hand side of the analyser.
  - 6. Collect, review and collate data

**Total Analysis Time:** 10 mins x 4 = 40 mins in morning 10 mins x 4 = 40 mins in afternoon plus preparation time

#### **Data Analysis**

The between-day precision of the Allegro be assessed by calculating the % coefficient of variation (%CV) from the mean and standard deviation from the replicate measurements. Acceptability criteria are determined by the medical director and/or institution. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1, 2].

#### **Data Review**



Appendix 2

**Between-Day Precision Study Data Collection Sheet** 

| Hospital | Name: | | | Dat | e of Stud | y: | | | _ | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System | Operator(s): | | | | | | | | | | | | |
| Referen | Reference Analyzer | | | | | | | | | | | | |
| Level 1 | Total Cholesterol, | Triglycerid | es and HDI | L Cholest | erol | | | | | | | | |
| Reference<br>Afterno<br>Reference<br>Reference | ce Analyzer Resul <sup>.</sup><br>ce Analyzer Resul <sup>.</sup><br>ce Analyzer Resul <sup>.</sup> | t mg/dL or<br>t mg/dL or<br>t mg/dL or<br>t mg/dL or | mmol/L Tr<br>mmol/L HI<br>mmol/L To<br>mmol/L Tr | iglyceride<br>DL Choles<br>otal Chole<br>iglyceride | es<br>esterol<br>esterol | | - | | | | | | |
| | System Name | | | | | | | | | | | | |
| | System Serial # | | | | | | | | | | | | |
| | Cartridge Lot # | | | | | | | | | | | | |
| Low QC<br>High QC | Range: | | | | | | | | | | | | |
| Tilgii QC | italige. | | Morni | ing | | | | | Afterno | on | | | |
| | Replicate # | Total Chol<br>mg/dL or<br>mmol/L | Total Chol<br>mg/dL or<br>mmol/L) | Trigs<br>mg/dL<br>or<br>mmol/L | Trigs<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | Total Chol<br>mg/dL or<br>mmol/L | Total Chol<br>mg/dL or<br>mmol/L) | Trigs<br>mg/dL<br>or<br>mmol/L | Trigs<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dl<br>or<br>mmol/ |
| | Day 1 | | | | | | | | | | | | |
| | Day 2 | | | | | | | | | | | | |
| | Day 3 | | | | | | | | | | | | |
| | Day 4 | | | | | | | | | | | | |
| | Day 5 | | | | | | | | | | | | |
| | Day 6 | | | | | | | | | | | | |
| | Day 7 | | | | | | | | | | | | |
| | Day 8 | | | | | | | | | | | | |
| | Day 9<br>Day 10 | | | | | | | | | | | <del> </del> | |
| Level 2 | Total Cholesterol, | irigiycerid | es and HDI | Lonolest | eroi | | | | | | | | |

Reference Analyzer Result mg/dL or mmol/L Total Cholesterol \_\_\_\_

| Reference Analyzer Result mg/dL or mmol/L Triglycerides |
|-------------------------------------------------------------|
| Reference Analyzer Result mg/dL or mmol/L HDL Cholesterol |
| <u>Afternoon</u> |
| Reference Analyzer Result mg/dL or mmol/L Total Cholesterol |
| Reference Analyzer Result mg/dL or mmol/L Triglycerides |
| Reference Analyzer Result mg/dL or mmol/L HDL Cholesterol |

| | System Name | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | | | | | |
| | Cartridge Lot # | | | | | | | | | | | | |
| Low QC | Range: | | | | | | | | | | | | |
| High QC | Range: | | | | | | | | | | | | |
| | | | Morn | ing | | | | | After | noon | | | |
| | Replicate # | Total Chol mg/dL or mmol/L | Total<br>Chol<br>mg/dL or<br>mmol/L) | Trigs<br>mg/dL<br>or<br>mmol/L | Trigs<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | Total<br>Chol<br>mg/dL or<br>mmol/L | Total<br>Chol<br>mg/dL<br>or<br>mmol/L) | Trigs<br>mg/dL or<br>mmol/L | Trigs<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L | HDL<br>Chol<br>mg/dL<br>or<br>mmol/L |
| | Day 1 | | | | | | | | | | | | |
| | Day 2 | | | | | | | | | | | | |
| | Day 3 | | | | | | | | | | | | |
| | Day 4 | | | | | | | | | | | | |
| | Day 5 | | | | | | | | | | | | |
| | Day 6 | | | | | | | | | | | | |
| | Day 7 | | | | | | | | | | | | |
| | Day 8 | | | | | | | | | | | | |
| | Day 9 | | | | | | | | | | | | |
| | Day 10 | | | | | | | | | _ | | _ | _ |

| 3. Total Cholesterol, Triglyceride and HDL Cholesterol |
|---|
| III. Method Comparison Study Protocol |
| Protocol based on the following guidance documents: |
| Clinical & Laboratory Standards Institute (CLSI). Method Comparison and Bias Estimation Using Patient Samples Approved Guideline – Second Edition. EP9-A2. |

#### **Purpose**

This protocol is designed to investigate how Allegro results compare to a recognized central laboratory reference method. These studies are important in order to establish the relationship between the Allegro System and the reference method with respect to statistical correlation and measurement bias. This protocol is designed and recommended for the Allegro System.

#### **Background**

Good practice dictates that the performance of medical devices such as the Allegro System be verified before the conductance of clinical studies. Verification studies include: method comparisons to determine how the results of the Allegro Systems compare to a recognized reference method, studies of imprecision to determine the reproducibility of the various tests available on the Allegro studies to determine the analytical trueness of the Allegro measurements. The protocol below describes how to conduct a method comparison (Allegro vs. Reference Method).

#### **Materials Needed**

- Nova Biomedical Allegro
- Allegro Lipid Cartridges
- Nova Biomedical Allegro Lipid Quality Control (QC) Solution
- Reference Analyzer and reagents
- 2mL plastic microcentrifuge tubes for decanting Na heparin or Li heparin samples
- Plastic 2mL disposable pipettes
- Full range of adjustable pipettes and tips
- If required appropriate Spiking stock solutions

#### **Important Factors to Consider**

Tests: Total Cholesterol, Triglycerides, HDL Cholesterol

Sample Type: Subject to change but to date:

- Capillary whole blood (from finger stick)
- Venous whole blood with anticoagulants Na heparin; Li heparin
- Venous plasma with anticoagulants Na heparin; Li heparin
- Serum

Sample Size: 5 µL

Time per Lipid: 10 mins

Linear Range of Operation for Total Cholesterol: 100-450 mg/dL (2.59-11.64 mmol/L)

**Linear Range of Operation for Triglyceride:** 50-600 mg/dL (0.56-6.76 mmol/L) **Linear Range of Operation for HDL Cholesterol:** 20-100 mg/dL (0.52- 2.59 mmol/L)

Please note that all parameters are processed at the same time.

#### **Normal Values:**

**Total Cholesterol:** Desirable is below 200 mg/dL (<5.17 mmol/L) **Triglycerides:** Desirable is below 150 mg/dL (<1.69 mmol/L) **HDL Cholesterol:** Desirable is 60 mg/dL and above (> 1.55 mg/dL)

#### **Control Levels:**

The Allegro supports two levels of controls. The following are suggested ranges for each parameter and level:

| | <b>Total Cholesterol</b> | Triglycerides | HDL Cholesterol |
|---|---|---|---|
| Low Level Target: | ~ 170 mg/dL | ~150 mg/dL | ~40 mg/dL |
| | (~4.40 mmol/L) | (~1.69 mmol/L) | (~1.04 mmol/L) |
| High Level Target: | ~ 240 mg/dL | ~300 mg/dL | ~60 mg/dL (1.55 mmol/L) |
| | (~6.21 mmol/L) | (~3.39 mmol/L) | (~1.55 mmol/L) |

#### **Procedure**

- 1. Fill out the requested information (Allegro serial numbers, cartridge lot numbers, QC lot numbers, QC ranges) on the provided Data Sheets (see Appendix).
- Perform quality control runs on the Allegro being evaluated and the reference analyzer. Record the results for all systems on the Data Sheet and make sure the results are within the manufacturer's control range. Proceed with testing only if all control results are within range.
- 3. 40-50 freshly collected/discarded whole blood venous, Na or Lithium heparin samples should be selected, that if possible, cover the analytical range across all analytes. Again spiking with appropriate spiking solutions may be required to completely cover the analytical range.
- 4. Ensure adequate mixing before analysis.
- 5. Analyse all samples in duplicate on the Allegro.
- 6. Samples should be spun down promptly (plasma) and then be analysed on the reference analyser.
- 7. Cartridges are stored at 4° each cartridge the lipids cartridge is only stable at RT for 1 hour
- 8. Run all samples in duplicate Allegro, the Lipids cartridge can only be run in the 660nm channel which is on the left hand side of the analyser.
- 9. Collect, Review and collate data.
- 10. Total Analysis Time: 10 mins  $\times$  80-100 = 800-1000 mins. Approx. 13.3 16.6 hrs plus preparation time
- 11. To reduce analysis time consider running samples in singles or perhaps less samples in duplicate whichever best suits site

#### **Data Analysis**

As part of this study paired total cholesterol, triglycerides and HDL cholesterol measurements will be collected. Analysis of accuracy is based on pairing individual results from the Allegro with the corresponding reference analyser measurement and calculating the difference (bias). Scatter plots and linear regression analysis are appropriate tools to assess the relationship between the Allegro results and the reference analyzer. Moreover, Bland-Altman plots can be used to assess the bias relative to the range of urine creatinine and urine Albumin concentrations studied. Investigators are referred to organizations such as CLSI and the International Standards Organization (ISO) which offer published acceptance criteria [1, 2]. The validity of the conclusions is dependent on experimental design, chiefly number of samples, the distribution of results, and the calibration of the reference analyzer.

#### **Data Review**

This data will be summarized in a summary report which will also include an assessment of precision. This report should be reviewed and signed off by the study site principal investigator. Results of this laboratory evaluation can be used to document verification of the Allegro System performance prior to the conductance of clinical studies.

#### References

1. Clinical & Laboratory Standards Institute (CLSI). *Method Comparison and Bias Estimation Using Patient Samples; Approved Guideline – Second Edition. EP9-A2.* 

## Appendix 4

## **Method Comparison Data Collection Sheet (Case Report Form)**


| Study Site: | Date of Study: |
|---------------------------------------------|-------------------|
| System Operator(s): | |
| Specimen Type (Na or Lithium heparin venou: | s blood) |
| Reference Analyzer Result mg/dL or mmol/L 1 | Total Cholesterol |
| Reference Analyzer Result mg/dL or mmol/L 1 | Friglycerides |
| Reference Analyzer Result mg/dL or mmol/L H | HDL Cholesterol |

| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial | | | | | | | | |
| | # | | | | | | | | |
| | Cartridge Lot # | | | | | | | | |
| Low QC | Range: | | | | | | | | |
| High QC | Range: | | | | | | | | |
| Specimen ID | Total Chol<br>mg/dL or<br>mmol/L | Total Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Total<br>Chol (mg/dL<br>or mmol/L) | Trigs<br>mg/dL or<br>mmol/L | Trigs<br>mg/dL/ or<br>mmol/L | Reference<br>Analyzer<br>Result Trig<br>(mg/dL or<br>mmol/L) | HDL Chol<br>mg/dL or<br>mmol/L | HDL Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result HDL<br>Chol(mg/dL<br>or mmol/L) |
| 1 | | | | | | | | | |
| 2 | | | | | | | | | |
| 3 | | | | | | | | | |
| 4 | | | | | | | | | |
| 5 | | | | | | | | | |
| 6 | | | | | | | | | |
| 7 | | | | | | | | | |
| 8 | | | | | | | | | |
| 9 | | | | | | | | | |
| 10 | | | | | | | | | |
| 11 | | | | | | | | | |
| 12 | | | | | | | | | |
| 13 | | | | | | | | | |
| 14 | | | | | | | | | |
| 15 | | | | | | | | | |
| 16 | | | | | | | | | |
| 17 | | | | | | | | | |
| 18 | | | | | | | | | |
| 19 | | | | | | | | | |
| 20 | | | | | | | | | |
| 21 | | | | | | | | | |
| 22 | | | | | | | | | |
| 23 | | | | | | | | | |
| 24 | | | | | | | | | |
| 25 | | | | | | | | | |

| 26 |
|----|
| 27 |
| 28 |
| 29 |

## Method Comparison Data Collection Sheet (Case Report Form)


| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | |
| | Cart Lot # | | | | | | | | |
| Specimen ID | Total Chol<br>mg/dL or mmol/L | Total Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Total<br>Chol (mg/dL<br>or mmol/L) | Trigs<br>mg/dL or<br>mmol/L | Trigs<br>mg/dL/ or<br>mmol/L | Reference<br>Analyzer<br>Result Trig<br>(mg/dL or<br>mmol/L) | HDL Chol<br>mg/dL or<br>mmol/L | HDL Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result HDL<br>Chol(mg/dL or<br>mmol/L) |
| 30 | | | | | | | | | |
| 31 | | | | | | | | | |
| 32 | | | | | | | | | |
| 33 | | | | | | | | | |
| 34 | | | | | | | | | |
| 35 | | | | | | | | | |
| 36 | | | | | | | | | |
| 37 | | | | | | | | | |
| 38 | | | | | | | | | |
| 39 | | | | | | | | | |
| 40 | | | | | | | | | |
| 41 | | | | | | | | | |
| 42 | | | | | | | | | |
| 43 | | | | | | | | | |
| 44 | | | | | | | | | |
| 45 | | | | | | | | | |
| 46 | | | | | | | | | |
| 47 | | | | | | | | | |
| 48 | | | | | | | | | |
| 48 | | | | | | | | | |
| 49 | | | | | | | | | |
| 50 | | | | | | | | | |
| 51 | | | | | | | | | |
| 52 | | | | | | | | | |
| 53 | | | | | | | | | |
| 54 | | | | | | | | | |
| 55 | | | | | | | | | |
| 56 | | | | | | | | | |
| 57 | | | | | | | | | |
| 58 | | | | | | | | | |
| 59 | | | | | | | | | |
| 60 | | | | | | | | | |
| 61 | | | | | | | | | |
| 62 | | | | | | | | | |
| 63 | | | | | | | | | |
| 64 | | | | | | | | | |
| 65 | | | | | | | | | |

| 66 |
|----|
| 67 |
| 68 |
| 69 |

## Method Comparison Data Collection Sheet (Case Report Form)


| | System Name | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | System Serial # | | | | | | | | |
| | Cart Lot # | | | | | | | | |
| Specimen ID | Total Chol<br>mg/dL or mmol/L | Total Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result Total<br>Chol (mg/dL<br>or mmol/L) | Trigs<br>mg/dL or<br>mmol/L | Trigs<br>mg/dL/ or<br>mmol/L | Reference<br>Analyzer<br>Result Trig<br>(mg/dL or<br>mmol/L) | HDL Chol<br>mg/dL or<br>mmol/L | HDL Chol<br>mg/dL or<br>mmol/L | Reference<br>Analyzer<br>Result HDL<br>Chol(mg/dL or<br>mmol/L) |
| 70 | | | | | | | | | |
| 71 | | | | | | | | | |
| 72 | | | | | | | | | |
| 73 | | | | | | | | | |
| 74 | | | | | | | | | |
| 75 | | | | | | | | | |
| 76 | | | | | | | | | |
| 77 | | | | | | | | | |
| 78 | | | | | | | | | |
| 79 | | | | | | | | | |
| 80 | | | | | | | | | |
| 81 | | | | | | | | | |
| 82 | | | | | | | | | |
| 83 | | | | | | | | | |
| 84 | | | | | | | | | |
| 85 | | | | | | | | | |
| 86 | | | | | | | | | |
| 87 | | | | | | | | | |
| 88 | | | | | | | | | |
| 89 | | | | | | | | | |
| 90 | | | | | | | | | |
| 91 | | | | | | | | | |
| 92 | | | | | | | | | |
| 93 | | | | | | | | | |
| 94 | | | | | | | | | |
| 95 | | | | | | | | | |
| 96 | | | | | | | | | |
| 97 | | | | | | | | | |
| 98 | | | | | | | | | |
| 99 | | | | | | | | | |
| 100 | | | | | | | | | |

| Name of Person Collecting Data: |
|--------------------------------------|
| Signature of Person Collecting Data: |
| Date: |

3. Total Cholesterol, Triglyceride and HDL Cholesterol
Summary Report Template

## **Total Cholesterol, Triglyceride and HDL Cholesterol Summary Report**

| Date: |
|----------------|
| Report Author: |
| Study Site: |
| · |

## Study Site Principal Investigator/Department:

**Materials and Methods** 

See Protocols I-IV. Any deviations from protocol should be noted here.

## **Summary of Results**

#### I. Precision Studies

Table 1. Total Cholesterol Within-Day Precision for Allegro

| | Low<br>Cholesterol | Mid<br>Cholesterol | High<br>Cholesterol |
|---|---|---|---|
| Mean mg/dL or mmol/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 2. Triglyceride Within-Day Precision for Allegro

| | Low<br>Triglyceride | Mid<br>Triglyceride | High<br>Triglyceride |
|---|---|---|---|
| Mean mg/dL or mmol/L | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 3. HDL Cholesterol Within-Day Precision for Allegro

| | Low<br>Cholesterol | Mid<br>Cholesterol | High<br>Cholesterol |
|---|---|---|---|
| Mean (mg/dL) | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 4. Total Cholesterol Between-Day Precision for Allegro

| | Low<br>Cholesterol | Mid<br>Cholesterol | High<br>Cholesterol |
|---|---|---|---|
| Mean (mg/dL) | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 5. Triglyceride Between-Day Precision for Allegro

| | Low<br>Triglyceride | Mid<br>Triglyceride | High<br>Triglyceride |
|---|---|---|---|
| Mean (mg/dL) | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

Table 6. HDL Cholesterol Between-Day Precision for Allegro

| | Low HDL<br>Chol | Mid HDL<br>Chol | High HDL<br>Chol |
|--------------------|-----------------|-----------------|------------------|
| Mean (mg/dL) | | | |
| Standard Deviation | | | |
| %CV | | | |
| N | | | |
| Matrix | | | |

## **III. Method Comparison**

Table 11. **Summary of Linear Regression Analysis Result**s: Total Cholesterol, Triglycerides and HDL Cholesterol for Allegro

| | <b>Total Cholesterol</b> | Triglyceride | HDL Cholesterol |
|---|---|---|---|
| Slope | | | |
| y-intercept (mg/dL) | | | |
| R <sup>2</sup> | | | |
| N | | | |
| Total Cholesterol Range | | | |
| mg/dL or mmol/L | | | |
| Triglyceride Range | | | |
| mg/dL or mmol/L | | | |
| HDL Cholesterol | | | |
| mg/dL or mmol/L | | | |

Table 12. Summary of Bland-Altman Results

| | <b>Total Cholesterol</b> | Triglyceride | HDL Cholesterol |
|---|---|---|---|
| Mean Bias (mg/dL) | | | |
| 95% Limits of Agreement | | | |
| Lower | | | |
| Upper | | | |
| Total Cholesterol Range<br>mg/dL or mmol/L | | | |
| Triglyceride Range<br>mg/dL or mmol/L | | | |
| HDL Cholesterol mg/dL or mmol/L | | | |

| Summary Findings | |
|------------------------------------------------|------|
| Allegro demonstrated | |
| This report has been reviewed and approved by: | |
| Signature of Study Site Principal Investigator | Date |
| Signature of MASA Director | Date |